CLINICAL TRIAL: NCT03834246
Title: Prognostic Factors for Smoke Inhalation Injury in Patients Admitted to Intensive Care
Brief Title: Smoke Inhalation Injury in Patients Admitted to Intensive Care
Acronym: fumeintox
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: Cicit805
Record Dates: First submitted 2018-11-21; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-11

CONDITIONS: Smoke Inhalation Injury; Morality
Keywords: Prognostic Factors; intensive care unit
MeSH Terms: conditions — Smoke Inhalation Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many Studies have shown that the smoke-inhalation injury is responsible for a high mortality mainly related to the systemic effects of carbon monoxide and cyanide. Respiratory lesions induced by smoke inhalation, is one of predictive factors of mortality.

The aim of the study is to identify the clinical and epidemiological characteristics of smoke-inhalation injury and to identify prognostic factors among these patients .

DETAILED DESCRIPTION:
The study is a monocentric, retrospective, descriptive and analytical study , betwen december 1997 and september 2018 in intensive care unit of university of hospital.

All patients aged over 18 year and who had received a diagnosis of smoke- inhalation injury and were admitted to the ICU of Medical University Hospital , a referral center in Paris providing HBO therapy , were potentially eligible for inclusion in this investigation.

Criteria used for recommending HBO therapy to a patient with transient or prolonged unconsciousness, abnormal neurologic findings on physical examination.

Data were analyzed to identify independent factors that may influence mortality.

ELIGIBILITY:
Inclusion Criteria

* Men or women over the age of 18
* Hyperbaric oxygen therapy between 1997 and 2018

Exclusion Criteria

* Patients under 18 years old.
* Patient opposed to the use of his data
* Patients not treated with hyperbaric oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We performed a retrospective study of patients admitted to a university affiliated hospital ICU between December 1997 and september 2018 following smoke -inhalation poisoning. Outcomes were survival to ICU discharge .
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 20 years
  survival study for the search of prognostic factors

SECONDARY OUTCOMES:
epidemiologic characteritics | 20 years
  description of quantitative and qualitative data

CONTACTS AND LOCATIONS:
Overall Officials: Rania BOUNAB, dr, Principal Investigator — Raymond Poincaré Hospital
Locations (1):
- Raymond Poincaré, Garches, France

REFERENCES:
- [Background] You K, Yang HT, Kym D, Yoon J, HaejunYim, Cho YS, Hur J, Chun W, Kim JH. Inhalation injury in burn patients: establishing the link between diagnosis and prognosis. Burns. 2014 Dec;40(8):1470-5. doi: 10.1016/j.burns.2014.09.015. Epub 2014 Oct 16. PMID 25406889
- [Background] Kim Y, Kym D, Hur J, Yoon J, Yim H, Cho YS, Chun W. Does inhalation injury predict mortality in burns patients or require redefinition? PLoS One. 2017 Sep 27;12(9):e0185195. doi: 10.1371/journal.pone.0185195. eCollection 2017. PMID 28953914
- [Background] Darling GE, Keresteci MA, Ibanez D, Pugash RA, Peters WJ, Neligan PC. Pulmonary complications in inhalation injuries with associated cutaneous burn. J Trauma. 1996 Jan;40(1):83-9. doi: 10.1097/00005373-199601000-00016. PMID 8577005
- [Background] Liao WC, Cheng WC, Wu BR, Chen WC, Chen CY, Chen CH, Tu CY, Hsia TC. Outcome and prognostic factors of patients treated in the intensive care unit for carbon monoxide poisoning. J Formos Med Assoc. 2019 Apr;118(4):821-827. doi: 10.1016/j.jfma.2018.09.005. Epub 2018 Oct 5. PMID 30293927
- [Background] Raphael JC, Annane D, Chevret S. Hyperbaric oxygen for acute carbon monoxide poisoning. N Engl J Med. 2003 Feb 6;348(6):557-60; author reply 557-60. No abstract available. PMID 12572578